CLINICAL TRIAL: NCT00541060
Title: Study of Factors of Genetic Susceptibility Associated to Severe Caries Phenotype in Young Patients. First Approach by Systematic Screening of Candidate Genes
Brief Title: Study of Factors of Genetic Susceptibility Associated to Severe Caries Phenotype
Acronym: Cariogene
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Aurélie GUIMFACK, Department of Clinical Research of developpement
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: P061009
Record Dates: First submitted 2007-10-04; First posted 2007-10-08 (Estimated); Last update posted 2010-12-20 (Estimated); Status verified 2010-11

CONDITIONS: Dental Caries
Keywords: caries susceptibility,enamel matrix,candidate genes,mutation
MeSH Terms: conditions — Dental Caries | interventions — Mutation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): 250 young patients presenting several carious lesions
  Interventions: Genetic: mutation
- B (Placebo Comparator): 160 young adults totally caries free
  Interventions: Genetic: mutation

INTERVENTIONS:
Genetic: mutation — a mutation of a gene coding
  Other Names: a mutation of a gene coding

SUMMARY:
Alteration of the post- eruptive enamel microstructure due to a mutation of a gene coding for a matrix protein could increase the susceptibility of the enamel to caries after tooth eruption. To identify in young patients with severe caries incidence, the occurrence of mutations in several candidate genes which result in an alteration of the enamel microstructure that could explain the high caries susceptibility of the patient.

DETAILED DESCRIPTION:
Although its prevalence has decreased dramatically in European countries, dental caries remains a burden for the society and especially for certain groups of the population. For example, 80% of the carious lesions are diagnosed in about 20% of the children. For years, the aetiology of this disease has been mainly related to environmental factors but recent data support the possibility of a human genetic contribution. Alteration of the post- eruptive enamel microstructure due to a mutation of a gene coding for a matrix protein could increase the susceptibility of the enamel to caries after tooth eruption. The main objective of this study will be to identify in young patients with severe caries incidence, the occurrence of mutations in several candidate genes which result in an alteration of the enamel microstructure that could explain the high caries susceptibility of the patient. With this aim, we will carry out a case- control multicentre European study on 250 young patients presenting several carious lesions and 160 young adults totally caries free. Patients with systemic or enamel pathologies such as amelogenesis imperfecta will not be included in the study. The study will consist of 2 visits, 1: inclusion and genetic test based on a salivary sample and 2: after 6 months, communication of the genetic test result to the patient and his parents. The main evaluation criteria will be the finding of a mutation on the candidates genes not resulting in an amelogenesis imperfecta phenotype but associated to a severe caries phenotype. If a direct relation between a mutation and a severe caries phenotype was shown, all the classical approaches, prevention protocols and treatments of caries would need to be reconsidered.

ELIGIBILITY:
Inclusion Criteria:

* Patients : presenting at least 3 active carious lesions aged 2 to 16 years old, written informed consent
* Volunteers : young adults 18 to 30 years old totally caries free

Exclusion Criteria:

* patients with systemic or enamel pathologies such as amelogenesis imperfecta
* osteogenesis imperfecta
* hypophosphatemia
* hypodermal dysplasia
* syndrome of Prader Willi
* Fluoroses
* toxic enamel dysplasia
* pregnancy or breast-feeding
* HYPOSIALORRHEA
* immunodepression status
* chronicle diseases
* anorexia or bulimia

Ages: 2 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 390 (Actual)
Dates: Start 2007-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
the finding of a mutation on the candidates genes not resulting in an amelogenesis imperfecta phenotype but associated to a severe caries phenotype | baseline, 6 months

SECONDARY OUTCOMES:
If a direct relation between a mutation and a severe caries phenotype was shown, all the classical approaches, prevention protocols and treatments of caries would need to be reconsidered. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Miller, MCU-PH, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Bretonneau, Paris, France